CLINICAL TRIAL: NCT01589081
Title: Effects of Progesterone on IV Nicotine-Induced Changes in Hormones and Subjective Ratings of Stimulant Drug Effect
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical studies never started; funding not received.
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Lukas, Director, Alcohol and Drug Abuse Research Center & Professor of Psychology (Neuroscience), Harvard Medical School, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2008-p-000454
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2013-01

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Female Smokers (Luteal Phase) (Active Comparator)
  Interventions: Drug: Intravenous Nicotine; Drug: Progesterone
- Female Smokers (Follicular Phase) (Active Comparator)
  Interventions: Drug: Intravenous Nicotine; Drug: Progesterone

INTERVENTIONS:
Drug: Intravenous Nicotine — Subjects will be given an IV challenge dose of nicotine or placebo in a constant volume of 2 mL on any study session day. The nicotine solutions (1.0 mg/70kg or 1.5 mg/70kg or 2.0 mg/70kg) will be administered over 1 min. This rate of drug delivery (2 mL over one minute) has been safe in our IRB-approved studies of nicotine. Most investigators have administered nicotine over 10 seconds without any adverse reactions. We concur with the IRB recommendation that the lower doses (1.0 mg/70kg; and 1.5 mg/70kg) will be administered first and the higher dose (2.0 mg/70kg) will be administered last.
  Other Names: IV Nicotine
Drug: Progesterone — To stimulate the luteal phase of the menstrual cycle, Prometrium capsules containing 200 mg of micronized progesterone or placebo (lactose containing) capsules will be administered orally at 120 minutes before the injection of IV nicotine.

SUMMARY:
The proposed clinical studies will analyze the interactions between progesterone, nicotine, alterations in endocrine hormones, mood and cardiovascular measures. It is hypothesized that the administration of progesterone at a dose that mimics luteal phase levels in normal cycling women will diminish the positive subjective effects of nicotine, as has been consistently observed for cocaine. This novel approach could have direct implications for facilitating smoking cessation treatment in women of reproductive age

DETAILED DESCRIPTION:
These clinical studies are designed to examine the effects of progesterone on IV nicotine induced changes on anterior pituitary (ACTH, LH, and Prolactin) and adrenal hormones (DHEA and cortisol). We also plan to study norepinephrine (NE) and epinephrine (E), because nicotine stimulates rapid release of NE and E in preclinical and clinical studies. The study will examine the acute effects of progesterone on the effects of IV nicotine on the HPG axis. Progesterone's influence on the acute effects of nicotine on the gonadal steroid hormones (estradiol, testosterone, progesterone) are unknown. The effects of progesterone on nicotine induced changes on gonadal steroid hormones and the reciprocal feedback regulation by LH will also be examined. The temporal covariance of progesterone influenced hormonal changes with serum nicotine levels and nicotine-induced changes in subjective states and cardiovascular measures will be analyzed. Finally, the covariance between the effects of progesterone on nicotine-induced changes in endocrine, subjective and cardiovascular effects and the temporal concordance with increases in serum nicotine and cotinine levels will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 40 who currently smoke at least 15 cigarettes every day, and who fulfill DSM-IV diagnostic criteria for nicotine dependence will be eligible for participation.
* No evidence of clinically significant disease based upon complete medical history and physical examination supervised by Dr. Arthur Siegel (Chief of Internal Medicine).
* Absence of DSM-IV Axis I Disorders other than nicotine dependence (305.10) as measured by the Structured Clinical Interview (SCID).
* Routine laboratory blood tests including complete blood count, electrolytes, BUN and creatinine, liver function tests, hepatitis panel and urinalysis will be performed. Laboratory parameters must be within the normal range. HBsAg must be negative but subjects who have hepatitis serology consistent with previous exposure to Hepatitis A, Hepatitis B, or Hepatitis C, but who do not have clinical and biochemical evidence of acute infection, will be acceptable.
* Hematocrit levels ≥ 35% for females.
* Serum pregnancy test (hCG beta subunit) results must be negative within 24 hrs of the study session day.
* Normal EKG.
* A Body Mass Index (BMI-ratio of weight (W) to height (H) squared; W/H2=kg/m2) of between 18.0 and 27.0 for women.
* Subjects must be able to read and understand instructions, as well as provide a valid informed consent.

Exclusion Criteria:

* Participants with any lifetime DSM-IV Axis I disorder other than nicotine dependence.
* Participants with clinically significant medical disorders.
* Women who are pregnant as determined by laboratory testing for serum beta hCG.
* Women who use hormonal contraceptive medications will not be accepted, because this would confound the hormonal measures.
* Women with a mean BMI of outside the range 18.0-27.0.
* Subjects with peanut/peanut oil allergies will be excluded.
* Participants diagnosed with lactose intolerance will be excluded.
* Participants who describe themselves as seeking treatment will not be selected but will be referred to local smoking cessation programs.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Effects of Progesterone on IV nicotine hormones and mood | From baseline to study completion (approximately 1 year)
  We are examining the effects of progesterone on IV nicotine induced changes in serum/plasma hormone levels and subjective states, as measured by a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Mello, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Alcohol and Drug Abuse Research Center at McLean Hospital, Belmont, Massachusetts, United States